CLINICAL TRIAL: NCT06238375
Title: Protocol for The Lipid Registry of Africa (LIPRA)
Brief Title: Protocol for The Lipid Registry of Africa
Status: Not yet recruiting | Type: Observational
Sponsor: European Atherosclerosis Society (Other)
Responsible Party: Sponsor
Other Study IDs: 3000124
Record Dates: First submitted 2024-01-24; First posted 2024-02-02 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: Acute Coronary Syndrome; Atherosclerosis
Keywords: Lipid Registry of Africa; Acute Coronary Syndrome; Cardiovascular Risk Factors; Multinational Study
MeSH Terms: conditions — Acute Coronary Syndrome; Atherosclerosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Premature Acute Coronary Syndrome (ACS) Patients in Africa: This cohort includes individuals diagnosed with premature Acute Coronary Syndrome (ACS), including subtypes like unstable angina, non-ST-segment elevation myocardial infarction (NSTEMI), and myocardial infarction with persistent ST-segment elevation (STEMI). These participants are under 55 years (men) or 65 years (women) and have been admitted to various cardiac facilities in Africa (Urban and rural) due to ACS-related symptoms.

SUMMARY:
The Lipid Registry of Africa (LIPRA) aims to understand why some individuals in Africa experience heart issues at a younger age than others. The study investigates factors causing heart problems in younger adults, particularly acute coronary syndrome (ACS). Acute coronary syndrome (ACS) includes various heart conditions like unstable angina and heart attacks. Researchers from multiple African countries collaborate to gather information from hospitals across the region. They focus on patients under 55 years (men) or 65 years (women) with heart issues.

Additionally, the study wants to compare different groups-men and women, urban and rural residents-to see if there are specific differences in how heart problems develop among them.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with premature Acute Coronary Syndrome (ACS) within the defined age range (≤55 years in men and ≤65 years in women).
* Patients admitted to designated cardiac facilities in Africa (Urban and rural).
* Diagnosed cases of ST-elevation myocardial infarction (STEMI) or non-ST-elevation myocardial infarction/unstable angina pectoris (NSTEMI/UAP) based on predetermined criteria including symptoms, electrocardiogram (ECG) alterations, and biomarker levels.
* Patients exhibiting an increase (above the 95th percentile) or decrease in serum troponin levels as per admission standards.

Exclusion Criteria:

* Individuals outside the defined age range for premature Acute Coronary Syndrome (ACS) diagnosis.
* Patients not admitted to designated cardiac facilities in Africa.
* Diagnosed cases not meeting the specified criteria for Acute Coronary Syndrome (ACS) subtypes (STEMI, NSTEMI/UAP) based on symptoms, electrocardiogram (ECG), and biomarker levels.

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The Lipid Registry of Africa (LIPRA) focuses on individuals residing in Africa (Urban and rural) diagnosed with premature Acute Coronary Syndrome (ACS). This encompasses patients admitted to specialized cardiac facilities in these regions meeting stringent criteria for ACS subtypes-ST-elevation myocardial infarction (STEMI) and non-ST-elevation myocardial infarction/unstable angina pectoris (NSTEMI/UAP). Inclusion mandates symptoms, electrocardiogram (ECG) alterations, and biomarker levels consistent with Acute Coronary Syndrome (ACS) within the specified age range (≤55 years in men, ≤65 years in women). The study aims to scrutinize the risk factor profile and demographics, uncovering the prevalence and impact of established and emerging risk factors for coronary artery disease. LIPRA, a multinational initiative, collaborates across diverse healthcare facilities, pooling data from multiple African countries.
Sampling Method: Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2024-04-30 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Risk factors prevalence | Through study completion, an average of 1 year
  The prevalence of traditional Cardiovascular (CV) risk factors among African patients with premature Acute Coronary Syndrome (ACS).

SECONDARY OUTCOMES:
Gender Difference in Risk Factors | Through study completion, an average of 1 year
  This secondary outcome aims to assess and compare the risk factor profiles between male and female individuals diagnosed with premature acute coronary syndrome (ACS) in Africa.
Prevalence of Familial Hypercholesterolemia (FH) According to the Dutch Lipid Clinic Network Score (DLCNS) | Through study completion, an average of 1 year
  This secondary outcome aims to determine the prevalence of Familial Hypercholesterolemia (FH) within the study population using the Dutch Lipid Clinic Network Score (DLCNS).
  The DLCNS is a diagnostic tool used to estimate the likelihood of FH based on a combination of genetic, clinical, and family history criteria. It assigns points across various categories, and the total score categorizes the probability of FH as "Definite," "Probable," "Possible," or "Unlikely." Minimum and Maximum Values: The DLCNS has a scoring system that ranges from 0 to >8 points. The minimum score (0 points) would typically indicate a lower likelihood of FH, while the maximum (>8 points) suggests a definite FH diagnosis.
Prevalence of the Use of Invasive Strategy Compared to Conservative Strategy for Managing Patients with Acute Coronary Syndrome (ACS) in Africa | Through study completion, an average of 1 year
  This secondary outcome aims to investigate the prevalence of the use of invasive strategy (e.g., coronary angiography and revascularization) compared to conservative strategy (medical management without immediate invasive procedures) for managing patients diagnosed with acute coronary syndrome (ACS) in Africa.

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf Reda, MD, Principal Investigator — The Egyptian Association of Vascular biology and Atherosclerosis (EAVA); Alexandros D. Tselepis, MD, PhD, Principal Investigator — Biochemistry-Clinical Chemistry, Chemistry Department, University of Ioannina, Greece; Alberto Zambon, MD, PhD, Principal Investigator — Department of Medicine -University of Padua School of Medicine - Italy; Alexander R.M. Lyons, PhD, Principal Investigator — Imperial College, London, Faculty of Medicine, School of Public Health

IPD SHARING:
Plan to Share IPD: Yes
The study protocol will be made available upon a reasonable request to the director of the project
Supporting Information: Study Protocol
Time Frame: One year after the end of the study.